CLINICAL TRIAL: NCT06360796
Title: A Phase I Study to Investigate the Absorption, Metabolism, Excretion, and Safety of [(14)C]ADC189 in Healthy Chinese Male Volunteers
Brief Title: Study of Pharmacokinetics and Metabolism on [(14)C]ADC189
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiaxing AnDiCon Biotech Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-ADC189-I-010
Record Dates: First submitted 2024-04-03; First posted 2024-04-11 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-03

CONDITIONS: Pharmacokinetics; Metabolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ADC189 (Experimental): 45 mg (about 100 μCi) [(14)C]ADC189
  Interventions: Drug: [(14)C]ADC189

INTERVENTIONS:
Drug: [(14)C]ADC189 — Each subject take a single oral dose of about 45 mg (about 100 μCi) [(14)C]ADC189 on Day 1 of the study, and be observed by 504 hours.

SUMMARY:
This study is designed to determined the metabolism, excretion, and substance balance of almonertinib of ADC189. The pharmacokinetic characteristics and safety profile of ADC189 was investigated following a single oral dose (45 mg/100 µCi) in healthy Chinese male participants.

DETAILED DESCRIPTION:
This study adopted a single-center, open, non-randomized, single-dose design. Six to eight healthy Chinese male subjects were planned to be enrolled, and the final aim is to collect all required samples and data from at least 6 subjects.

After each subject take a single oral dose of 45 mg (about 100 μCi) [14C]ADC189 on Day 1, whole blood, plasma, urine and feces samples were collected at specified time points during the study. The total radioactivity was measured to calculate the ratio of total radioactivity of whole blood to total radioactivity of plasma, pharmacokinetic parameters, recovery rate and excretion pathway data of total radioactivity in whole blood and plasma. Meanwhile, the radioactive metabolite spectrum and structural identification of main metabolites in plasma, urine and feces were performed to obtain the pathway and characteristics of main metabolic elimination of ADC189 in human body, as well as circulating metabolites ≥10% of total radioactivity exposure in plasma.

ELIGIBILITY:
Inclusion Criteria:

* 1. healthy Chinese male subjects within 18 to 45 years old inclusive;
* 2. body weight over 50 Kg, and within a BMI range of 19.0 to 26.0 kg/m2 inclusive;
* 3. has no sperm donation plan, no family planning and voluntarily adopts strict contraceptive methods during the study period and within six months after the completion of the trial;
* 4. able to comprehend and willing to sign an Informed Consent Form (ICF).

Exclusion Criteria:

* 1. history or presence of an abnormal ECG;
* 2. participation in more than 1 other radiolabeled investigational study drug trial within 12 months prior to Check-in;
* 3. exposure to significant radiation within 12 months prior to Check-in;
* 4. participation in any other investigational study drug trial;
* 5. use of any prescription medications/products within 14 days prior to Check-in;
* 6. use of any drug that affects drug metabolism enzymes or transporters (P-gp and BCRP) in the 30 days prior to taking the study drug, as detailed in Appendix 5;
* 7. receipt of blood products within 1 month prior to Check-in.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2023-11-24 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
The Area Under the Curve (AUC) of [(14)C]ADC189 and its metabolites | 504 hours
The Maximum Plasma Concentration [Cmax] of [(14)C]ADC189 and its metabolites | 504 hours
The whole blood and serum concentrations of total radioactivity of [(14)C]ADC189 (about 100 μCi) | 504 hours
The urinary and fecal recovery of total radioactivity of [(14)C]ADC189 (about 100 μCi) | 504 hours

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affilicated Hospital of Bengbu Medical University, Bengbu, Anhui, China

IPD SHARING:
Plan to Share IPD: No